CLINICAL TRIAL: NCT04197011
Title: Investigating the Effects of Micro-processor Controlled Knee Components on the Function and Performance of Individuals With Transfemoral Amputation
Brief Title: Advanced Prosthetic Devices for Lower Limb Amputees
Status: Completed | Type: Observational
Sponsor: Nottingham Trent University (Other)
Responsible Party: Principal Investigator, Dr. Cleveland T. Barnett, Principal Investigator, Nottingham Trent University
Other Study IDs: IRAS237030
Record Dates: First submitted 2019-12-05; First posted 2019-12-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Prostheses and Implants
Keywords: Prosthetics; Microprocessor; Hydraulic
MeSH Terms: interventions — Artificial Limbs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prosthesis users: Individuals with unilateral transfemoral amputation.
  Interventions: Device: prosthetic device
- Control: Individuals without unilateral transfemoral amputation.

INTERVENTIONS:
Device: prosthetic device — Individuals with TFA will use a combination of prosthetic devices.
  Groups: Prosthesis users

SUMMARY:
Lower limb amputation is an emerging global health concern. Currently, there are over 1.6 million amputees in the U.S. and around 6000 new amputations are recorded per annum in the UK. These numbers are expected to double by 2050 due to the increasing aging population and the adverse health issues such as diabetes, representing a significant, growing problem in western society. A lower limb amputation results in the loss of the biological joint structures such as the ankle and knee, along with the associated musculature. In order to overcome these physical losses, many lower limb amputees are provided with a prosthetic limb that enable them to participate in activities of daily living. The design and function of these prosthetic limbs varies widely, with some being very basic, non-articulating, semi-rigid structures while other more advanced components are computer controlled or incorporate robotic function. Lower limb amputees have been shown to fall more often when compared to age matched individuals without lower limb amputation. This has been reported to be partly a result of a less stable walking pattern. Given that the prosthetic limb provided and it's functional capability is a large component of how well a lower limb amputee is able to walk, it is important to understand what the effects of and potential benefits are from using more advanced prosthetic devices, such as micro-processor controlled knee joints and articulating ankle joints.

Therefore, the aim of the current study is to investigate the effects of combining more advanced prosthetic ankle-foot and knee components on the biomechanics of activities of daily living in individuals with above knee amputation.

DETAILED DESCRIPTION:
Study Background Lower limb amputation is an emerging global health concern. Currently, there are over 1.6 million amputees in the U.S. and around 6000 new amputations are recorded per annum in the UK. These numbers are expected to double by 2050 due to the increasing aging population and the adverse health issues such as diabetes, representing a significant, growing problem in western society. A lower limb amputation results in the loss of the biological joint structures such as the ankle and knee, along with the associated musculature. In order to overcome these physical losses, many lower limb amputees are provided with a prosthetic limb that enable them to participate in activities of daily living. The design and function of these prosthetic limbs varies widely, with some being very basic non-articulating semi-rigid structures while other more advanced components are computer controlled and function robotically. Advanced ankle components have been shown to provide lower limb amputees with a number of benefits including increased walking speed, improved symmetry between legs and increased forward progression. In addition, micro-processor controlled knee components, recently made available through the NHS via NHS England Clinical commissioning, have shown a number of benefits. These benefits are stated as being '…enhanced stability and stumble recovery, which improves fall management and reduces the incidence of falls. This supports the increases in self-reported improved individual mobility and independence. MPKs also improve controlled sitting and standing, walking gait symmetry, stair decent, controlled step over step descent down a slope, reduced energy expenditure, and given different modes for different activities an ability to manage obstacles more easily'. Given that the prosthetic limb provided and their functional capability is a large component of how well a lower limb amputee is able to walk, it is important to understand what the effects of and potential benefits are from using more advanced prosthetic devices, such as micro-processor controlled knee joints. Also, as these components are used in conjunction with ankle-foot devices, it is important to know what the optimal combination may be to gain the most benefits from both prosthetic components.

Study Aim The aim of the current study is to investigate the effects of combining more advanced prosthetic ankle-foot and knee components on the biomechanics of activities of daily living in individuals with above knee amputation.

ELIGIBILITY:
Inclusion Criteria:

1. Transfemoral amputation: Individuals who have had unilateral transfemoral amputation.
2. Demographics: Adult, community-dwelling individuals above the age of 18 in order to provide written informed consent for themselves.
3. Mental Capacity: Ability to comprehend and understand communication and instruction in English in order to consent and safely participate in study as assessed verbally.
4. Mobility level: Prospective participants must be able to negotiate obstacles such as ramps and stairs thus displaying a level of mobility commensurate with a medicare K3 functional classification level.
5. Endurance Capacity: Able to walk continuously for periods of up to two minutes at a time in order to complete the clinical walking tests.
6. Vision: Good (corrected) vision to safely walk in well-lit areas.
7. Cardiovascular Health: No self-reported unresolved cardiovascular complaints to avoid any cardiovascular complications when performing activities of daily living.
8. Able to travel: Data collection will take place at Nottingham Trent University, Clifton Campus.

For the otherwise healthy control (CTRL) group, the same criteria apply, with the exception of those pertaining specifically to amputation status.

Exclusion Criteria:

1. Pain: Experience undue musculo-skeletal pain during walking that causes individual to stop and not be able to continue when walking at a self-selected speed.
2. Disease/Illness: Unable and/or unsafe to carry out tasks due to disease/illness such as rheumatoid arthritis.
3. Injury: Current neuromuscular, musculoskeletal injury.
4. Falls: Falls regularly (>1 a month) as determined using the PROFANE fall definition. Excludes recreational, sporting or occupational falls outside of this definition.
5. Residuum health: Presence of significant blisters, wounds and rash which prevent prosthesis, sock and liner to be worn comfortably.
6. Residuum stability: Observing substantial changes to the physical condition of the lower limb that requires medical attention as judged by the participant, and if after consenting and participating in the study, individuals are referred to mobility services due to a degradation of the physical condition of either lower limb.
7. Unable to follow instruction or cognitive deficits: Risk of further injury whilst completing tasks incorrectly.
8. Not able to understand written and verbal English: All communication will be in English as the University does not provide translation services.
9. For the otherwise healthy control (CTRL) group, the same criteria apply, with the exception of those pertaining specifically to amputation status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study aims to recruit two groups of participants, one group of individuals with unilateral transfemoral amputation (TFA) and a group of otherwise healthy control participants (CRTL). Both groups are required to satisfy inclusion and exclusion criteria and provide written informed consent in order to participate.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Obstacle Course Completion Time (seconds) | All experimental conditions - up to six weeks
  The total time taken to complete one lap of a custom walking course in seconds.

SECONDARY OUTCOMES:
Two-minute walk (2MWT) test (metres) | All experimental conditions - up to six weeks
  The total distance walked in two minutes along a 13m walkway.
The timed up and Go (TUG) test | All experimental conditions - up to six weeks
  Assessment of mobility, where participants are timed whilst rising from an arm chair, walking three metres, and returning to a sitting position on the chair
The L-test | All experimental conditions - up to six weeks
  This is a modified version of the TUG test, where individuals rise from a chair, walk three metres, turn 90 degrees, walk seven metres, turn 180 degrees, walk seven metres, turn 90 and return to a sitting position in the same chair.
Berg Balance Scale | All experimental conditions - up to six weeks
  Grading the participants' ability to perform a number of functional tasks such as moving from standing to sitting which are scored on a five point scale from zero (worst) to four (best).
EQ-5D-5L | All experimental conditions - up to six weeks. Only applicable for participants who are currently trialling an MPK.
  Standardised measure of health related quality of life which is used internationally. A visual analogue scale requires participants to rate their health on a zero (worst) to 100 (best) scale.
Activities Balance Confidence Scale-UK (ABC-UK) | All experimental conditions - up to six weeks. Only applicable for participants who are currently trialling an MPK.
  A self-report, quality of life outcome measure, relating balance confidence to functional activities. Scores are reported from zero (worst) to 100 (best) in terms of their confidence in completing a particular task.
Locomotor Capabilities Index (LCI) | All experimental conditions - up to six weeks. Only applicable for participants who are currently trialling an MPK.
  Assessment of self-perceived capability to perform 14 different locomotor activities when using a prosthesis. This is rated on a five point scale from zero (worst) to four (best).
The Houghton Scale | All experimental conditions - up to six weeks. Only applicable for participants who are currently trialling an MPK.
  A 4-item instrument that assesses prosthetic use in and reflects a person's perception of prosthetic use. This is rated on a four point scale from zero (worst) to three (best).
Custom Falls Report | All experimental conditions - up to six weeks. Only applicable for participants who are currently trialling an MPK.
  A recall on the incidence and circumstances around falls experienced which are reported every 30 days.
The Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form | All experimental conditions - up to six weeks. Only applicable for participants who are currently trialling an MPK.
  Taking pain related aspects of this survey to quantify self-reported pain issues in prosthesis users. For example, pain interference when completing a task is rated on a five point scale from 'not at all' (best) to 'very much'.

CONTACTS AND LOCATIONS:
Overall Officials: Cleveland Barnett, Ph.D, Principal Investigator — Nottingham Trent University
Locations (1):
- The Biomechanics Lab, CELS Building, Nottingham Trent University, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided